CLINICAL TRIAL: NCT01035801
Title: An OpenLabel, Multicenter, Non-randomized, ActiveControlled, SingleDose Escalation, Study to Evaluate the Pharmacodynamics,Pharmacokinetics,Safety, and Tolerability of IN-105 Under Fed Conditions In Patients With Type 1 Diabetes Mellitus
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral Insulin (IN-105) in Type 1 Diabetes Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was temporarily paused due to an unanticipated bioanalytical issue.
Sponsor: Biocon Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN105-CT1-005-09
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Indium-105; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IN105 (Experimental): Prandial Oral Insulin
  Interventions: Drug: IN-105
- Insulin Lispro Injection (Active Comparator)
  Interventions: Drug: Insulin Lispro Injection

INTERVENTIONS:
Drug: IN-105 — Prandial Oral Insulin
  Arms: IN105
Drug: Insulin Lispro Injection — Insulin Lispro Injection
  Arms: Insulin Lispro Injection

SUMMARY:
The purpose of this study is to see whether IN-105 (oral insulin) is able to control increase in blood glucose after eating a meal. This study will also tell whether single tablet of IN-105 is safe for patients with Type 1 diabetes mellitus who are currently taking insulin injections.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 18-45 years inclusive
2. Established diagnosis of T1DM for at least 1-year
3. Body mass index of 18.5-29.9 kg/m2 inclusive
4. Stable weight with no more than 5 kg gain or loss within 3 months of screening
5. HbA1c ≤ 8.0%
6. On stable insulin or an insulin analogue regimen for at least 3 months

Exclusion Criteria:

1. Any hypersensitivity or allergy
2. Positive urine ketones test at screening visit.
3. ECG abnormality
4. total daily insulin >1 IU/kg and/or >0.7 IU/Kg of basal insulin and/or >0.6 IU/Kg of prandial insulin.
5. Patient with a clinically significant abnormality
6. Evidence of severe secondary complications of diabetes
7. History of drug or alcohol dependence or abuse
8. Patients currently on systemic or inhaled glucocorticoids or other drugs, which may affect glycemic control.
9. Patients treated with blood-glucose lowering drugs other than insulin or insulin analogues in the last 4 weeks prior to screening or during the study
10. History of two or more severe episodes of hypoglycemia (defined by ADA criteria) within 6 months prior to screening and/or patients with history of low blood glucose level episodes suggestive of hypoglycemia unawareness (loss of warning symptoms of hypoglycemia). Investigator to assess this criterion based on the subject filled questionnaire.
11. Any hospitalization or emergency room visit due to poor diabetes control within 6 months prior to screening.
12. Impaired hepatic function (ALT or AST value greater than 2 X Upper limit of reference range and/or serum bilirubin ≥1.5 X Upper limit of reference range at the screening visit).
13. Impaired renal function (serum creatinine ≥1.5 X Upper limit of reference range at screening).
14. Hemoglobinopathies, haemolytic anaemia, anaemia of chronic disease, or any factor affecting the measurement of HbA1c.
15. Any electively planned surgery requiring hospitalization during the study period.
16. Pregnancy, lactation, or planned pregnancy during the study duration.
17. The patient has received another investigational drug within 6 weeks prior to screening
18. Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08-21 (Actual); Primary Completion 2011-03-12 (Actual); Study Completion 2011-03-12 (Actual)

PRIMARY OUTCOMES:
AUC (Insulin and Blood Glucose) | 0-130 min

SECONDARY OUTCOMES:
AUC (Insulin and Blood Glucose) | 0-70 min, 0-190 min and 0-250 min
Frequency of Adverse Events | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. K.M. Prasanna Kumar, MD, DM, Principal Investigator — CEO and Consultant Endocrinologist, Bangalore Diabetes Hospital, #16/M, Miller tank Bed Area, Thimmaiah Road, Vasanthnagar, Bangalore-560052; Dr. Aravind R Sosale, DNB, Principal Investigator — Director, Diacon Hospital,Diabetes Care and Research Centre, 359-360, 19th Main, Ist Block,Rajajinagar,Bangalore-560010.; Dr. Sanjay Kalra, MD, DM, Principal Investigator — Bharti Research Institute of Diabetes & Endocrinology (BRIDE), Bharti Hospital, Wazir Chand Colony, Kunjpura, karnal, Hariyana- 132001; Dr Bipin Kumar Sethi, MD, DM, Principal Investigator — Care Hospital, Road 1, Banjara Hills, Hyderabad - 500034; Dr. Neeta Deshpande, MD, Principal Investigator — Belgaum Diabetic Centre, Ground floor,Beside mahila Vastu Bhander, Maruti Gali, Belgaum- 590001
Locations (5):
- India (5):
  - Care Hospital, Hyderabad, Andhra Pradesh
  - Bharti Research Institute of Diabetes and Endocrinology, Karnāl, Haryana
  - Diacon Hospital,(Diabetes Care and Research Centre), Bangalore, Karnataka
  - Bangalore Diabetes Hospital, Bangalore, Karnataka
  - Belgaum Diabetic Centre, Belagavi, Karnataka